CLINICAL TRIAL: NCT06345196
Title: The Effect of Motivational Interviewing on Well-being, Stress and Difficulties in Individuals With Diabetes
Brief Title: Motivational Interviewing Applied to Individuals With Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Betül Bal, Lecturer, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BozokUni
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Motivational Interviewing; Stress; Well-Being, Psychological; Diabetes Mellitus; Type2diabetes
MeSH Terms: conditions — Psychological Well-Being; Diabetes Mellitus | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): Motivational interviewing will be conducted in four sessions and the session duration will be maximum 40 minutes. The session will be conducted individually and online once a week. For the individual interview, the appropriate day and time will be determined with the individuals with diabetes and the researcher before the first session and the sessions will continue on the same day and time every week. The researcher will remind the participant about the time of the session by calling the participant by phone one day before each session. Motivational interview sessions will be held online on the Whatsapp platform.
  Interventions: Behavioral: motivational interview
- Control (No Intervention): The patients in the control group, on the other hand, did not undergo any intervention other than their routine treatment and care. The patients were followed for four weeks. Before the study, data collection tools were applied to the patients. Again, after the study started and the study ended, all other data collection tools were applied, except the "Patient Information Form".

INTERVENTIONS:
Behavioral: motivational interview — Motivational interviewing will be conducted in four sessions and the session duration will be maximum 40 minutes. The session will be conducted individually and online once a week. For the individual interview, the appropriate day and time will be determined with the individuals with diabetes and the researcher before the first session and the sessions will continue on the same day and time every week. The researcher will remind the participant about the time of the session by calling the participant by phone one day before each session. Motivational interview sessions will be held online on the Whatsapp platform.
  Arms: Motivational Interviewing

SUMMARY:
This study will be conducted using a randomized controlled trial design to evaluate the effect of online individual motivational interviewing on well-being, stress and difficulties in individuals with diabetes. The study will be conducted between March 2024 and March 2025 with individuals with Type 2 Diabetes who are followed up in Yozgat Bozok University Health Practice and Research Center Internal Medicine Polyclinic. The motivational interview group will receive a motivational interview once a week, lasting a maximum of 40 minutes, consisting of a total of four sessions. Chi-square (X2), t-test, repeated measures analysis of variance, Pearson correlation coefficient, partial eta-square and linear regression analysis will be used to evaluate the data.

DETAILED DESCRIPTION:
Approximately 537 million people worldwide have diabetes and it is estimated to reach 643 million in 2030 and 783 million in 2045. In this context, the prevalence of diabetes is increasing and 1.5 million people die each year due to diabetes. Diabetes is a chronic disease that requires complex care activities and multiple decision-making related to self-management. In particular, the most common is type 2 diabetes in adults, which occurs when the body becomes resistant to insulin or does not produce enough insulin. Daily self-management of the disease is necessary for individuals with type 2 diabetes to achieve healthy glucose levels, minimize the effects of the disease on their daily lives and reduce the risk of developing complications. The main elements of self-management in individuals with diabetes include taking medication, maintaining a healthy diet, regular physical activity, foot care and monitoring blood glucose for insulin users.

Managing diabetes is a process that requires continuous effort and adherence to multiple health behaviors, and many patients have difficulty managing this chronic condition. This situation increases stress in individuals and causes deterioration in well-being and psychosocial status.

Stress in individuals with diabetes can negatively affect problem-solving skills and lead to poor self-management behavior. However, it has also been reported that positive well-being in individuals with diabetes has a good effect on disease management (better glucose control, reduced disease burden, increased work productivity and reduced mortality). However, individuals with type 2 diabetes have been found to have lower well-being than the general population. Therefore, it is important to develop stress coping strategies and support positive well-being for people with diabetes.

The control of diabetes depends on the individual's healthy lifestyle behaviors and disease management as well as the pharmacological treatment option. However, many systematic reviews show that motivational interviewing is an effective intervention method in the treatment of diabetes. These studies have shown that it has positive effects on diet and weight management, diabetes self-management, medication adherence, and glycemic control in individuals with diabetes. Looking at the literature, although less stress and positive well-being are important to overcome the difficulties in disease management in individuals with diabetes, studies on supporting stress and positive well-being in type 2 diabetes patients are limited. In this context, this study will be conducted to determine the effect of motivational interviewing applied to individuals with diabetes on well-being, stress and difficulties.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study,
* Having a diagnosis of Type 2 Diabetes,
* HbA1C values outside the normal range for the last 2-3 months.

Exclusion Criteria:

* Having a diagnosis of Type 1 Diabetes,
* Having limitations in reading and understanding Turkish.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in coping with stress | 4 weeks
  This scale will be administered twice before and after the intervention to determine the patients' coping methods with stress. The scale consists of three sub-dimensions: problem-focused coping (8 items), social support-focused coping (7 items) and avoidance-focused coping (8 items). The scale consists of a total of 23 items, 20 of which are positively worded and three items (items 10, 17, 20) are negatively worded. A score of 23-115 can be obtained from the whole scale. The higher the score obtained from the whole scale and subscales reflects the tendency of the person to use the relevant ways of coping with stress.

SECONDARY OUTCOMES:
State of Well-Being Change | 4 weeks
  The scale consists of 5 items containing 5 positive statements about the participant's emotions in the last 2 weeks. Each item is evaluated on a 6-point Likert-type scale ranging from 0-5; a score of 0 indicates no positive emotions in the last 2 weeks, while a score of 5 indicates continuous positive emotions. Raw scores are converted into a scoring scale between 0-10. A score below 50 indicates low mood.

OTHER OUTCOMES:
Changing Strength and Difficulties in Diabetes | 4 weeks
  As a result of the factor analysis, the scale of strengths and difficulties in type 2 diabetes consisted of 3 sub-dimensions and 30 items in total. Each item in the scale is in 5-point Likert type and the minimum score that can be obtained from the scale is 30 and the maximum score is 150. There are no reverse items in the scale. An increase in the score obtained from the scale indicates that the difficulties experienced by individuals with type 2 diabetes increase.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Akdağmadeni School of Health, Yozgat
  - Bozok University, Yozgat